CLINICAL TRIAL: NCT00245115
Title: Ex Vivo Expansion of Mafosfamide Purged CD34+ Cells in Patients With Acute Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Expiration of study supply
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0563 CDR0000453619; P01CA070970 (NIH); P30CA006973 (NIH); NCT00246649 (obsolete NCT alias)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Leukemia
Keywords: adult acute myeloblastic leukemia without maturation (M1); childhood acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); childhood acute myeloblastic leukemia with maturation (M2); adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3); adult acute myelomonocytic leukemia (M4); childhood acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); childhood acute monoblastic leukemia (M5a); childhood acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); childhood acute erythroleukemia (M6); adult acute megakaryoblastic leukemia (M7); childhood acute megakaryocytic leukemia (M7); adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); secondary acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Promyelocytic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Congenital Abnormalities | interventions — Filgrastim; Busulfan; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Procedure: in vitro-treated bone marrow transplantation
Procedure: in vitro-treated peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving colony-stimulating factors, such as G-CSF, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected. Treating stem cells collected from the patient's blood or bone marrow with chemotherapy in the laboratory removes any remaining cancer cells. Chemotherapy or radiation therapy is given to the patient to prepare the bone marrow for stem cell transplant. The treated stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This clinical trial is studying how well an autologous peripheral stem cell or bone marrow transplant using laboratory-treated cells works in treating patients with acute leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of ex vivo expanded mafosfamide-purged CD34-positive cells for autologous peripheral blood stem cell or bone marrow transplantation in patients with acute leukemia.
* Determine the duration of aplasia associated with the use of ex vivo cytokine expanded mafosfamide-purged cells in patients treated with this regimen.
* Determine, preliminarily, the event-free survival of patients treated with this regimen.

OUTLINE: This is a pilot study.

* Mobilization and stem cell collection: Patients receive cyclophosphamide IV and filgrastim (G-CSF) subcutaneously (SC) or IV once daily for 7-14 days followed by leukapheresis to collect peripheral blood stem cells (PBSCs). Some patients may also undergo bone marrow (BM) harvest if sufficient PBSCs are not collected. Patients with a sufficient number of stem cells or BM (5 x 10^6 PBSC/kg or 3 x 10^8 BM cells/kg) proceed to autologous PBSC transplantation (PBSCT) or BM transplantation (BMT).
* CD34-positive cell selection and mafosfamide purging: Collected PBSCs and/or BM are treated in the laboratory to isolate CD34-positive cells. A minimum of 1 x 10^6 nucleated CD34-positive BM cells/kg or 2 x 10^6 nucleated CD34-positive PBSCs/kg must be available after selection to proceed to mafosfamide-purging. The selected cells are then treated in vitro with mafosfamide to purge remaining leukemic cells. One third of the mafosfamide-purged cells are then cryopreserved for future use and 2/3 of the mafosfamide-purged cells proceed to ex vivo expansion.
* Ex vivo expansion: The remaining CD34-positive mafosfamide-purged cells are treated in vitro with stem cell factor, G-CSF, and recombinant human thrombopoietin and incubated for 12-14 days.
* Myeloablative therapy: Patients receive busulfan on days -9 to -6 and cyclophosphamide on days -5 to -2.
* PBSCT or BMT: Patients undergo autologous PBSCT or BMT using CD34-positive mafosfamide-purged cryopreserved cells and ex vivo expanded CD34-positive mafosfamide-purged cells on day 0 followed by G-CSF SC or IV once daily until blood counts recover.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute leukemia meeting 1 of the following criteria:

  * High-risk acute myeloid leukemia (AML) in first complete remission (CR) with no matched family donor available, including any of the following types:

    * Secondary AML
    * AML with chromosome 5 or 7 abnormalities
    * AML with trisomy 8
    * AML with 6;9 chromosomal translocation
    * AML with 11q23 chromosomal abnormality
    * AML with multiple or complex chromosomal abnormalities
    * AML with FAB M6 or M7
  * AML in second CR (CR2) with no eligible HLA-identical sibling donor available
  * High-risk acute lymphoblastic leukemia (ALL) with no eligible HLA-identical sibling donor available, including any of the following types:

    * Philadelphia chromosome-positive ALL
    * ALL with 11q23 chromosomal abnormality
    * ALL in CR2
* Eligible for and willing to undergo bone marrow transplantation
* No intermediate- or good-risk acute leukemia in CR1

Exclusion Criteria

* Availability of a suitable matched HLA-identical sibling marrow donor
* Intermediate or good risk acute leukemia in CR1 (39)
* Age greater than 70
* Weight less than 10 kg
* Any risk of pregnancy - all female patients must have an effective form of contraception or be infertile due to hysterectomy, fallopian tube, surgery or premature menopause.
* HIV Infection: Patients must be HIV negative for inclusion.
* Poor organ function as defined in the BMT Policies and Procedures Manual.

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Number of patients infused with Mf-treated cells with successful expansion | 2 weeks
  Number of patients with successful expansion of a CD34 selected, mafosfamide purged autograft.

SECONDARY OUTCOMES:
Duration of aplasia as determined by Number of Days to Absolute Neutrophil Count (ANC) recovery | 1 month
Event free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: B. Douglas Smith, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No